CLINICAL TRIAL: NCT05838261
Title: Prospective Evaluation of Speech Function Through Patient- and Parent-response Outcome Measurements Following Surgical Treatment of Velopharyngeal Insufficiency in Children With Isolated or Combined Cleft Palate
Brief Title: Prospective Evaluation of Speech Function Through Patient- and Parent-response Outcome Measurements in Velopharyngeal Insufficiency
Status: Recruiting | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Karolinska University Hospital (Other); Uppsala University Hospital (Other); University Hospital, Linkoeping (Other); Skane University Hospital (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Rebecka Wiberg, Principal Investigator, Umeå University
Other Study IDs: 2023-VPI-RWiberg
Record Dates: First submitted 2023-03-29; First posted 2023-05-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Velopharyngeal Insufficiency in Children With Isolated or Combined Cleft Palate
Keywords: Velopharyngeal insufficiency; Pharyngeal flap; Patient- and parent-reported outcome measurements; Cleft palate
MeSH Terms: conditions — Velopharyngeal Insufficiency; Cleft Palate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with cleft palate with velopharyngeal insufficiency undergoing surgical treatment: Children with combined or isolated cleft palate with velopharyngeal insufficiency undergoing surgical treatment with pharyngeal flap
  Interventions: Procedure: Pharyngeal flap

INTERVENTIONS:
Procedure: Pharyngeal flap — Children with combined or isolated cleft palate with velopharyngeal insufficiency undergoing surgical treatment with pharyngeal flap will be evaluated with patient- and parent reported outcome measures before and after the surgery.

SUMMARY:
Cleft lip and/or palate (CL/P) is the most common congenital malformation, with about one in 500 children born with CL/P in Sweden, corresponding to approximately 175 births annually. Depending on the extent of the cleft palate, the degree of functional loss varies, but both eating, hearing, speech, bite and appearance can be affected.

Patients treated for isolated or combined cleft palate may suffer from velopharyngeal insufficiency (VPI), which means difficulties in closing the passage between the oral and nasal cavities during speech. Velopharyngeal insufficiency is associated with hypernasality, audible nasal air leakage and weak articulation, which might lead to difficulties with communication and social stigmatization.

The most common form of speech-improving surgery is a posterior based velopharyngeal flap, creating a bridge between the palate and the posterior pharyngeal wall to more easily compensate for the abnormal airflow through the nose during speech. However, surgical management of VPI is challenging, with variable success rates reported in the literature. In a retrospectively based questionnaire study on patients who underwent surgical treatment of VPI, 30% experienced only a small speech improvement or no improvement at all. In addition, postoperative speech impairment have also been reported, as well as perioperative bleeding and postoperative sleep apnea. Thus, selecting the patients who benefit most from speech-improving surgery is therefore of great importance.

The aim with the current study is evaluation of speech function through patient- and parent-response outcome measurements following surgical treatment of velopharyngeal insufficiency in children with isolated or combined cleft palate.

ELIGIBILITY:
Inclusion Criteria:

* All children < 18 years of age with isolated or combined cleft palate that will undergo pharyngeal flap surgery due to velopharyngeal insufficiency, as well as their parents, in any of the 6 specialized cleft center in Sweden.

Exclusion Criteria:

* Cognitive impairment making it difficult to understand the study.

Ages: 0 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: All children < 18 years with isolated or combined cleft palate undergoing surgical treatment of velopharyngeal insufficiency in any of the 6 specialized cleft centers in Sweden will be invited to the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Speech function | Change in speech function will be evaluated preoperatively and 1 year postoperatively
  Speech function will be evaluated through the patient response outcome measurement CLEFT-Q pre- and postoperatively. Each CLEFT-Q scale is transformed into scores that range from 0-100, with higher scores reflecting a better outcome.
Speech function | Change in speech function will be evaluated preoperatively and 1 year postoperatively.
  Speech function will be evaluated through the parent-response outcome measurement Intelligibility in Context Scale pre- and postoperatively. The maximum and minimum value ranges from 0-35 respectively, with higher scores reflecting a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Wiberg, MD PhD, Principal Investigator — Umeå University
Locations (6):
- Sweden (6):
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Skånes University Hospital, Malmo
  - Karolinska University Hospital, Stockholm
  - Plastic Surgery Unit, Umeå University hospital, Umeå
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No
This is a multicenter study so the other researchers will be part of analysing the data, however only on group level.